CLINICAL TRIAL: NCT05120557
Title: Evaluation of Diagnostic Performances of a New Point-of-care Ultrasound System for the Detection of Fibrotic NASH and the Assessment of Liver Disease Severity in Patients With Known or Suspected Chronic Liver Disease
Brief Title: Point-of-care Ultrasound Screening and Assessment of Chronic Liver Diseases and NASH
Acronym: POCUS-NASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: E-Scopics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ES211
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-04

CONDITIONS: Liver Diseases; Liver Cirrhosis; NASH - Nonalcoholic Steatohepatitis; Non-Alcoholic Fatty Liver Disease; Fibrosis, Liver; Steatosis of Liver
Keywords: Elastography; Ultrasound attenuation; Sound speed; Ultrasound
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis; Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Intervention Model Description: All patients recruited will receive routine care for liver assessment followed by an exam using the device subject of the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main arm (Experimental): Main study arm
  Interventions: Device: Ultrasound liver assessment

INTERVENTIONS:
Device: Ultrasound liver assessment — The intervention consists in an ultrasound exam performed with the ultrasound medical device subject of the research.
  Other Names: Elastography; Ultrasound attenuation; Sound speed

SUMMARY:
The main objective of the study is to determine the diagnostic performances of an ultraportable diagnostic ultrasound system for the assessment of liver fibrosis severity in patients with NASH, and to compare them to other non-invasive tests.

DETAILED DESCRIPTION:
This is a prospective cross-sectional study that will recruit approximately 1000 patients across 30 clinical sites in Europe and the USA.

The target recruited population will include adult patients at risk of, or with known chronic liver diseases, whether or not screened for inclusion in NASH pharmaceutical trials.

After being informed about the study objectives and potential risks, patients who consent to participate will undergo an non-invasive external ultrasound exam of their liver using an ultraportable diagnostic ultrasound system. The system will derive quantitative information related to physical and acoustic properties of the liver tissue, which are known to correlate with the severity of chronic diffuse liver diseases such as fibrosis and steatosis.

The study will also assess the repeatability, reproducibility and robustness of quantitative parameters. Collected data will also enable exploring ultrasound-based liver tissue characterization correlated to NASH-specific histological lesions such as intra-hepatic inflammation and hepatic cell ballooning.

ELIGIBILITY:
Inclusion Criteria:

* Any of the following criteria:

  * Patients with known chronic liver diseases referred to liver-specific exams by their referring physician as part of the routine practice, including a VCTE exam, with or without a blood test, a MRI/MRE exam, a liver biopsy,
  * Patients screened for fibrotic NASH in the context of NASH pharmaceutical trials, for which a data sharing agreement has been signed between E-Scopics and the pharmaceutical trial promoter,
* Patients who consent in written to participate in the Clinical Investigation after being orally informed on the objectives and methods of the Clinical Investigation,
* European patients covered by a social security program

Exclusion Criteria:

* Patients under 18 years of age or over 80 years of age,
* Patients with active implants such as pacemakers, defibrillators, pumps, etc.
* Patients presenting wounds at the location where the ES1 probe shall be placed on patients' skin,
* Adult patients under social tutorship, or unable to provide informed consent when not subject to tutorship measures,
* Pregnant and breastfeeding women,
* People deprived of their freedom rights
* People who have been hospitalized without giving informed consent or under emergency situation,
* People admitted in a social or sanitary institution for other reasons than the Clinical Investigation,
* Patients included in another research study that could interfere with the present Clinical Investigation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Elastography diagnostic performance | At study completion, 1 year
  Differences between areas under ROC curves for the ES1 liver stiffness measurement, used as a diagnostic measure of liver fibrosis severity, and other methods, in NASH patients.
Diagnostic performance estimates | At study completion, 1 year
  Estimates of diagnostic performances at a defined cutoff, for binary diagnostic objectives (detect ≥ F2, ≥ F3, or F4):
  1. Sensitivity, specificity, and diagnostic accuracy
  2. Positive and negative predictive values

SECONDARY OUTCOMES:
Liver stiffness robustness indicators | At study completion, 1 year
  1. Dispersion and standard deviation of measurements
  2. Intra-class Correlation Coefficients (ICC) and 95% confidence intervals for intra-operator repeatability
  3. Intra-class Correlation Coefficients (ICC) and 95% confidence intervals for inter-operator reproducibility
  4. Intra-subject variance
  5. Intra-operator variance
  6. Standard error on measurements
Equivalence with other methods | At study completion, 1 year
  1. R² correlation coefficient and p-value between ES1 and VCTE liver stiffness measurements
  2. R² correlation coefficient and p-value between ES1 and MRE liver stiffness measurements
  3. Average of quadratic errors between 2 equipment
  4. Concordance Correlation Coefficients (CCC) and 95% confidence intervals

OTHER OUTCOMES:
Exploratory outcome 1: Liver steatosis | At study completion, 1 year
  1. R² correlation coefficient and p-value between ES1 ultrasound attenuation measurements and MRI PDFF
  2. Concordance Correlation Coefficients (CCC) and 95% confidence intervals, and Bland-Altman graphs between ultrasound attenuation measurements and MRI PDFF
  3. R² correlation coefficient and p-value between ES1 speed of sound measurements and MRI PDFF
  4. Concordance Correlation Coefficients (CCC) and 95% confidence intervals, and Bland-Altman graphs between speed of sound measurements and MRI PDFF
Exploratory outcome 2: Intra-hepatic inflammation and/or hepatocytes ballooning | At study completion, 1 year
  1. Correlation coefficients between ES1 parameters or combinations of parameters and histological scoring for lobular inflammation (A0 to A3) and/or ballooning.
  2. If relevant, area under the ROC curve for combinations of ES1 parameters or combinations of parameters used as a diagnostic measures of liver inflammation severity using histological scoring for lobular inflammation (A0 to A3)
  3. If relevant for given binary diagnostic objectives (detect ≥ A1, ≥ A2, or A3), calculate optimal diagnostic cutoffs and estimate diagnostic performances
Exploratory outcome 3: Liver NAS Score | At study completion, 1 year
  1. Correlation coefficients between ES1 parameters or combinations of parameters and histological NAS score (NAS 0 to NAS 8).
  2. If relevant, area under the ROC curve for combinations of ES1 parameters or combinations of parameters used as a diagnostic measure of NAFLD-related activity using the histological NAS score (0 to 8)
  3. If relevant, for given binary diagnostic objectives (detect < NAS 3, ≥ NAS 3, ≥ NAS 5), calculate optimal diagnostic cutoffs and estimate diagnostic performances

IPD SHARING:
Plan to Share IPD: No